CLINICAL TRIAL: NCT03481036
Title: Direct Acting Antiviral Agent (DAA) Therapy Is Safe and Efficacious in Pediatric Patients With Chronic Hepatitis C: Real World Data From the Public Health Perspective
Brief Title: DAA Therapy in Pediatric Patients With Chronic Hepatitis C
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Directorate of Health and Family Welfare, Punjab (Other)
Responsible Party: Principal Investigator, Radha K Dhiman, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEC/2018/000323
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Chronic Hepatitis c
Keywords: Mukh Mantri Punjab Hepatitis C Relief Fund,MMPHCRF; Direct acting antiviral agents (DAA); Chronic Hepatitis C; Pediatric population; Adolescent Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non cirrhotic (Active Comparator): Sofosbuvir (SOF)+Daclatasvir (DCV) for 12 weeks Patients < 35 kg will be given half doses of medications and patients ≥35 kg will be given adult dosages of SOF (400 mg), LDV (90 mg) and DCV (60 mg) per day
  Interventions: Drug: Direct Acting Antivirals
- Genotype 1,4,5 and 6 with cirrhosis (Active Comparator): Sofosbuvir (SOF)+ Ledipasvir (LDV) for 12-weeks + weight based Ribavirin Patients < 35 kg will be given half doses of medications and patients ≥35 kg will be given adult dosages of SOF (400 mg) and LDV (90 mg) per day
  Interventions: Drug: DAAs in Cirrhotics Genotye 1,4,5,6
- Genotype 2 and 3 with Cirrhosis (Active Comparator): Sofosbuvir (SOF)+Daclatasvir (DCV) for 12 weeks+ weight based Ribavirin Patients < 35 kg will be given half doses of medications and patients ≥35 kg will be given adult dosages of SOF (400 mg) and DCV (60 mg) per day
  Interventions: Drug: DAAs in Cirrhotics Genotype 2/3

INTERVENTIONS:
Drug: Direct Acting Antivirals — Sofosbuvir and Daclatasvir
  Other Names: DAAs in Non Cirrhotics
  Arms: Non cirrhotic
Drug: DAAs in Cirrhotics Genotype 2/3 — Sofosbuvir and Daclatasvir with weight based ribavirin
  Arms: Genotype 2 and 3 with Cirrhosis
Drug: DAAs in Cirrhotics Genotye 1,4,5,6 — Sofosbuvir and Ledipasvir with weight based ribavirin
  Arms: Genotype 1,4,5 and 6 with cirrhosis

SUMMARY:
The Mukh-Mantri Punjab Hepatitis C Relief Fund (MMPHCRF) is a public health initiative for prevention and control of hepatitis C in the Punjab state, India. The efficacy of decentralised public health services and safety of 12- or 24-weeks of sofosbuvir (SOF) + ledipasvir (LDV) or SOF + daclatasvir (DCV) with or without ribavirin (RBV) in the treatment of pediatric chronic hepatitis C will be assessed

DETAILED DESCRIPTION:
Consecutive chronic hepatitis C (HCV) infected children [age: ≥12 to <18 years; both treatment-naïve (TN) and treatment-experienced, (TE)] are being enrolled.

Genotyping is not recommended for non-cirrhotic or TN patients and are treated with SOF+DCV for 12-weeks, while genotyping is recommended for patients with cirrhosis and TE patients.

Patients with liver cirrhosis or TE and genotype (GT)-3 are being treated with SOF+DCV for 24 weeks,

while non-GT-3 patients are being treated with SOF+LDV for 24-weeks. Patients < 35 kg are being given half doses of medications and patients ≥35 kg are being given adult dosages of SOF (400 mg), LDV (90 mg) and DCV (60 mg) per day.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C, all genotypes
* Ages eligible for study: ≥12 to <18 years (Child)
* Gender eligible for study: either
* Treatment-naive or treatment-experienced: either

Exclusion Criteria:

* Chronic liver disease of a non-HCV etiology
* serum creatinine >1.5 mg/dL
* Evidence of hepatocellular carcinoma or other malignancy
* Co-infection with hepatitis B virus, or HIV
* Significant cardiovascular, pulmonary, or neurological disease
* Evidence of a malabsorption syndrome that could interfere with absorption of orally administered medications
* History of solid organ or bone marrow transplantation.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06-18 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained Virological Response (SVR 12) | 12 weeks after completion of therapy
  HCV RNA undetectable by quantitative Real time Polymerase Chain Reaction (PCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dhiman RK, Grover GS, Premkumar M, Taneja S, Duseja A, Rathi S, Satsangi S. Direct-acting antiviral Therapy Is Safe and Effective in Pediatric Chronic Hepatitis C: The Public Health Perspective. J Pediatr Gastroenterol Nutr. 2019 Jan;68(1):74-80. doi: 10.1097/MPG.0000000000002139. PMID 30211847